CLINICAL TRIAL: NCT05818163
Title: Association of Perioperative Electroencephalography Spectral Analysis With Postoperative Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202208066DINA
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia; Pain; EEG
Keywords: electroencephalography spectral analysis; postoperative complications; anesthesia monitoring
MeSH Terms: conditions — Pain; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with postoperative complications: Patients who experience postoperative complications after anesthesia, with symptoms such as pain, nausea and vomiting, delirium, and agitation.
  Interventions: Device: electroencephalography spectral analysis
- without postoperative complications: Patients who do not experience postoperative complications after anesthesia, free from symptoms such as pain, nausea and vomiting, delirium, and agitation.
  Interventions: Device: electroencephalography spectral analysis

INTERVENTIONS:
Device: electroencephalography spectral analysis — Before inducing general anesthesia in the patient entering the operating room, an anesthesia depth monitoring patch is attached to the forehead, and EEG data during anesthesia is collected using the currently used anesthesia depth monitoring device.
  The EEG data is transformed into a frequency and energy distribution and density spectral array (DSA) graph using Fourier transform (FFT) for spectral analysis.
  Other Names: density spectral array; patient state index (PSI)

SUMMARY:
Using data from electroencephalogram (EEG) obtained through intraoperative depth of anesthesia monitoring devices, combined with clinical symptoms such as postoperative pain and delirium, investigate their correlation and verify whether intraoperative EEG spectral analysis can predict the occurrence of postoperative pain, nausea and vomiting, restlessness, or delirium in patients undergoing surgery.

DETAILED DESCRIPTION:
Due to the complexity of the original EEG waveforms, previous anesthesia depth monitoring systems only calculated a single index, such as Bispectral index (BIS) or patient state index (PSI), to determine the state under anesthesia. However, a single numerical change may not reflect the true state under anesthesia. By analyzing the original EEG waveforms, more information can be obtained, such as density spectral array (DSA) and power spectral density, which can quantify the energy distribution at various brain wave frequencies. This allows anesthesiologists to determine the effects of medication on brain waves and the effects of surgical stimulation on brain waves during surgery.

After obtaining the signed informed consent form, before inducing general anesthesia in the patient entering the operating room, an anesthesia depth monitoring patch is attached to the forehead, and EEG data during anesthesia is collected using the currently used anesthesia depth monitoring device. The monitoring process starts from the beginning of general anesthesia until the end of the surgery, and the EEG recording is stopped only when the patient wakes up from general anesthesia and leaves the operating room.

By using the original EEG during anesthesia depth monitoring to conduct spectral analysis and combining it with common post-anesthesia adverse symptoms such as pain, nausea and vomiting, delirium, and restlessness, a correlation analysis is conducted between the quantified EEG values and postoperative symptoms. This verifies whether intraoperative EEG spectral analysis can predict the occurrence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20 years or older.
2. Patients who received general anesthesia within the our hospital system.

Exclusion Criteria:

1. Individuals with suspected infections, such as a fever higher than 38.3℃
2. Individuals with renal dysfunction, such as those with creatinine levels higher than 1.5 or those who require long-term dialysis
3. Individuals with cardiac dysfunction, such as those with NYHA class III or higher heart failure or coronary heart disease Individuals with neurological diseases, such as those with brain tumors, dementia, stroke, or epilepsy
4. Vulnerable populations, such as minors (under 20 years of age), pregnant women and fetuses, prisoners, adults who cannot give informed consent, individuals with disabilities, individuals with mental illness, residents of nursing homes or long-term care facilities, or those who may be subject to coercion or unable to make decisions freely.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 20 years or older who received general anesthesia within the National Taiwan University Hospital system.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
pain in the postanesthesia care unit | up to 2 hours, postanesthesia
  Visual Analog Scale (VAS) > 3 in the postanesthesia care unit
agitation in the postanesthesia care unit | up to 2 hours, postanesthesia
  Richmond Agitation-Sedation Scale (RASS)>2 in the postanesthesia care unit

SECONDARY OUTCOMES:
delirium | up to 2 days, postanesthesia
  delirium after anesthesia, CAM-ICU
nausea and vomiting | up to 1 day, postanesthesia
  nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Cancer Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No